CLINICAL TRIAL: NCT02519205
Title: Measuring Fatigue in Triage: A Pilot Study
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00065707
Record Dates: First submitted 2015-08-05; First posted 2015-08-10 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-02

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ED Nurses: ED triage nurses from Duke University Hospital (DUH) and Duke Regional Hospitals (DRH).
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey
  Other Names: Karolinska Sleepiness Scale; Samn-Perelli Seven Point Fatigue Scale

SUMMARY:
The purpose of this study is to determine how the length of a triage shift (i.e. 4 vs., 8 vs., 12 hours) affects fatigue levels among triage nurses in the Emergency Department (ED).

DETAILED DESCRIPTION:
This will be a prospective descriptive pilot study. The demographic data forms and the adapted reaction questionnaires will be administered to subjects via pen and paper after obtaining informed consent at the conclusion of the staff meetings. They will be collected by administrative assistants and placed into a secure drop box, located in the study coordinator's office. Only the assigned unique subject ID will be used on all data forms.

During the ED triage data collection phase, administrative assistants will be on-site to give triage nurses the fatigue questionnaire. It will be completed using pen and paper every two hours, with subjects cued to complete the questionnaire by administrative assistants.

After the subject completes the survey, he/she will place it in an envelope and hand it to the administrative assistant who will place it into a secured drop box, located in a study coordinator's office. No PHI or identifying data will be on the completed surveys. Each participant will only use the previously assigned unique subject ID, known only to the study coordinator & Co-PIs, & PI. The key to the unique ID will be kept in a locked secure file accessible only by the study coordinator and Co-PI.

Data will be collected over a total of six 24-hour periods. The first 24-hour data collection period will take place on a high volume day (Monday) in which triage nurses will be assigned to 12-hour triage shifts. The second 24-hour data collection period will take place on a low volume day (Sunday) in which triages nurses will again be assigned to 12-hour triage shifts. The third 24-hour data collection period will take place on a high volume day (Monday) in which nurses will be assigned to 8-hour triage shifts. The fourth 24-hour data collection period will take place on a low volume day (Sunday) in which nurses will again be assigned to 8-hour triage shifts. The fifth 24-hour data collection period will take place on a high volume day (Monday) in which nurses will be assigned to 4-hour triage shifts. The sixth 24-hour data collection period will take place on a low volume day (Sunday) in which nurses will again be assigned to 4-hour triage shifts.

ELIGIBILITY:
Inclusion Criteria:

-Eligible nurses include those who:

* are regularly assigned to triage
* have demonstrated competency by passing the ESI Triage class. (Nurses in both emergency departments are required to attend a course in Emergency Severity Index (ESI), as well as demonstrate competency through ESI testing prior to being assigned to work in the triage area. Before taking the course, a nurse is required to have one year of nursing experience.)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ED Triage nurses
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2015-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Fatigue level, as measured by questionnaire | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Regional Hospital, Durham, North Carolina, United States